CLINICAL TRIAL: NCT06159673
Title: A Master Protocol for Three Independent, Seamlessly Enrolling, Double-blind, Placebo-controlled Efficacy and Safety Studies of ACP-204 in Adults With Alzheimer's Disease Psychosis
Brief Title: ACP-204 in Adults With Alzheimer's Disease Psychosis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-204-006
Record Dates: First submitted 2023-11-27; First posted 2023-12-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease Psychosis
Keywords: Alzheimer's disease psychosis; Hallucinations; Delusions
MeSH Terms: conditions — Hallucinations; Delusions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ACP-204 30 mg (Experimental): Administration once daily at approximately the same time of day, with or without food
  Interventions: Drug: ACP-204
- ACP-204 60 mg (Experimental): Administration once daily at approximately the same time of day, with or without food
  Interventions: Drug: ACP-204
- Placebo (Placebo Comparator): Administration once daily at approximately the same time of day, with or without food
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACP-204 — ACP-204 is a potent and selective antagonist/inverse agonist of 5-hydroxytryptamine (serotonin) receptor subtype 2A.
  Arms: ACP-204 30 mg; ACP-204 60 mg
Drug: Placebo — ACP-204 matching placebo
  Arms: Placebo

SUMMARY:
This is a master protocol for 3 independent, seamlessly enrolling, multicenter, randomized, double-blind, placebo-controlled, parallel-group studies in patients with ADP

* Substudy 1 (Phase 2) will evaluate efficacy and dose response of ACP-204 30 and 60 mg vs placebo. This substudy will be initiated first.
* Substudies 2A and 2B (both: Phase 3) will be confirmatory studies of either both doses (ACP-204 30 and 60 mg, respectively) or a single dose from Part 1 vs placebo. Substudies 2A and 2B will be performed independently of each other and will commence after enrollment of Part 1.

All 3 substudies will be analyzed independently of each other.

Each substudy individually will consist of a screening period (up to 49 days); a double-blind treatment period (6 weeks); a safety follow-up period (30 days) for patients not rolling over into an open-label extension study; and vital status follow-up (for patients who terminated their substudy early).

ELIGIBILITY:
Inclusion Criteria:

* Is male or female and ≥55 and ≤95 years of age living in the community or in an institutionalized setting
* Meets clinical criteria for possible or probable AD based on the 2011 National Institute on Aging-Alzheimer Association (NIA-AA) criteria
* Meets the revised criteria for psychosis in major or mild neurocognitive disorder established by the International Psychogeriatrics Association (IPA)
* Has either blood-based biomarker or documented evidence (e.g. positron emission tomography, cerebrospinal fluid biomarker) indicating amyloid plaque deposition and neuropathologic change consistent with AD
* Has a prior magnetic resonance imaging or computed tomography scan of the brain that is consistent with the diagnosis of AD
* Meets revised criteria for psychosis in major or mild neurocognitive disorder as per International Psychogeriatrics Association
* MMSE score ≥6 and ≤24
* Psychotic symptoms for at least 2 months
* Lives in a stable place of residence and there are no plans to change living arrangements
* Has a designated study partner/caregiver
* Able to complete all study visits with a study partner/caregiver
* Must be on a stable dose of cholinesterase inhibitor or memantine, if applicable

Exclusion Criteria:

* Requires treatment with a medication prohibited by the protocol
* Is in hospice and receiving end-of-life palliative care, or has become bedridden
* Requires skilled nursing care
* Psychotic symptoms that are primarily attributable to delirium, substance abuse, or a medical or psychiatric condition other than dementia
* Known history of cerebral amyloid angiopathy, epilepsy, central nervous system neoplasm, or unexplained syncope
* Atrial fibrillation
* Symptomatic orthostatic hypotension
* Protocol-defined exclusionary clinical laboratory findings
* Treatment with anti-tau therapy or donanemab within 2 months prior to Screening

Additional inclusion/exclusion criteria apply. Subjects will be evaluated at screening to ensure that all criteria for study participation are met.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1074 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Scale for the Assessment of Positive Symptoms-Hallucinations and Delusions subscales (SAPS-H+D) total score change from baseline (Substudies 1, 2A, 2B) | From baseline to Week 6
  The SAPS-H+D subscales are a measure of two psychotic symptoms: hallucinations and delusions. The SAPS-H+D total score is the sum of the scores of the Hallucinations and Delusions subscales. The hallucinations domain score (SAPS-H) is the sum of the 7 hallucinations item scores, and the delusions domain core (SAPS-D) is the sum of the 13 delusions item scores.

SECONDARY OUTCOMES:
Clinical Global Impression-Improvement in the ADP context (CGI-I-ADP) score | Week 6
  The CGI-I scale is a clinician-rated, 7-point scale used to rate the improvement in symptoms at the time of assessment, relative to the symptoms at Baseline. The CGI-I-ADP scale is the CGI-I scale applied in the ADP context, in which hallucinations and delusions are the symptoms of interest.

CONTACTS AND LOCATIONS:
Locations (142):
- United States (45):
  - Chandler Clinical Trials, Chandler, Arizona
  - Clinical Endpoint LLC, Scottsdale, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - ATP Clinical Research, Costa Mesa, California
  - Neuro-Pain Medical Center, Fresno, California
  - National Institute of Clinical Research, Garden Grove, California
  - Humanity Clinical Research Corp, Aventura, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - First Excellent Research Group, Doral, Florida
  - New Life Medical Research Center Inc., Hialeah, Florida
  - Reliable Clinical Research LLC., Hialeah, Florida
  - Homestead Associates in Research Inc., Miami, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Central Miami Medical Institute, Miami, Florida
  - Advanced Clinical Research Network, Corp, Miami, Florida
  - Verus Clinical Research, Miami, Florida
  - Future Care Solution, LLC, Miami, Florida
  - MediClear Medical & Research Center, Inc., Miami, Florida
  - ABBA Medical Group LLC, Miami, Florida
  - Visionary Investigators Network, Miami, Florida
  - Quantum Clinical Trials, Miami Beach, Florida
  - New Med Research, Miami Gardens, Florida
  - Floridian Neuroscience Institutue, Miami Lakes, Florida
  - Combined Research Orlando Phase I IV, Orlando, Florida
  - Psych Me Medical Research Inc, Tampa, Florida
  - Neuroscience Research Institute, West Palm Beach, Florida
  - Revive Research Institute, Inc., Elgin, Illinois
  - Grace Research, LLC, Shreveport, Louisiana
  - Khan Revive Research Institute, Rochester Hills, Michigan
  - Alivation Research, LLC, Lincoln, Nebraska
  - Dent Neurologic Institute, Amherst, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Regional Neurological Associates, The Bronx, New York
  - Insight Clinical Trials LLC, Beachwood, Ohio
  - Valley Medical Research, Centerville, Ohio
  - Abington Neurological Associates, Abington, Pennsylvania
  - Horizon Clinical Research Group, Cypress, Texas
  - Prolato Clinical Research Center-Patton, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Clinical Trial Network LLC, Houston, Texas
  - Kaleidoscope Clinical Research, Houston, Texas
  - Steven South Goldstein MD and Associates, Houston, Texas
  - World Research Link, Pasadena, Texas
  - R & H Clinical Research Inc., Stafford, Texas
  - Tranquil Clinical Research, Webster, Texas
- Brazil (13):
  - L2IP - Instituto de Pesquisas Clínicas Ltda, Brasília
  - Hospital Universitario de Brasilia, Brasília
  - TrialTech Tecnologia com Pesquisas em Medicamentos, Curitiba
  - Inst. de Neurologia de Curitiba Hospital Ecoville, Curitiba
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo
  - Hospital Moinhos de Vento, Porto Alegre
  - Nucleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Facili-Centro Integrado de Psiquiatria, São Bernardo do Campo
  - BR Trials-Ensaios Clinicos e Consultoria, São Paulo
  - Hospital Sao Paulo, São Paulo
  - Santa Paula Hospital Clinical Research Center, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina USP, São Paulo
- Bulgaria (12):
  - ET Dr. Ivo Natsov - AIPSMC in Psychiatry, Cherven Bryag
  - Medical Center Lifemed, Kardzhali
  - DCC "Higia", Pazardzhik
  - Medical center Medconsult Pleven OOD, Pleven
  - UMHAT Sv. Georgi EAD, Plovdiv
  - Medical center Spectar-Plovdic EOOD, Plovdiv
  - Mental Health Centre - Prof. N Shipkovenski EOOD, Sofia
  - DCC St. Vrach and St. St. Kuzma and Damian OOD, Sofia
  - UMHAT "Alexandrovska" EAD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Intermediea, Sofia
  - UMHAT Prof. Dr. St. Kirkovich AD, Stara Zagora
- Chile (4):
  - Psicomed Estudios Medicos, Antofagasta
  - Biomedica Research Group, Santiago
  - Especialidades Medicas L y S, Santiago
  - CIC de la Universidad Catolica CICUC, Santiago
- Czechia (8):
  - BRAIN-SOUL THERAPY s.r.o., Kladno, Czech Republic
  - Ad71 S.R.O., Prague, Czech Republic
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - NEUROHK s.r.o, Choceň
  - CLINTRIAL s.r.o., Prague
  - FORBELI s.r.o., Prague
  - INEP medical s.r.o, Prague
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- France (12):
  - Hopital Neurologique Bron, Bron
  - Centre pour Personnes Âgées, Colmar
  - Centre Memoire Ressources Recherche CMRR, Dijon
  - CHU de Limoges-Hopital Dupuytren, Limoges
  - Hospices Civils de Lyon HCL, Lyon
  - Hôpital Lariboisière, Paris
  - Hopital BROCA, Paris
  - CHU Rouen-Hospital Charles Nicolle, Rouen
  - Hopital Purpan, Toulouse
  - Hôpital La Grave, Toulouse
  - CHRU de Tours- Hopital Bretonneau, Tours
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Italy (10):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Neurologia-Fondazione Instituto G. Giglio, Cefalù
  - IRCCS Neuromed Istituto Neurologico Mediterraneo, Isernia
  - Ospedale San Raffaele, Milan
  - Fondazione Policlinico Uni Campus Bio-Medico di Roma, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - AOU Policlinico Umberto I, Roma
  - Azienda Ospedaliera Universitaria OO. RR. S., Salerno
  - Dipartimento di Neuroscienze Rita Levi Montalcini, Torino
  - Azienda Ospedaliera Card. G. Panico, Tricase
- Mexico (10):
  - Iecsi S.C., Monterrey, N.L
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Hospital Universitario Dr. Gonzalo Valdes Valdes, Coahuila
  - Clinical Research Institute S.C, Estado de México
  - Health Pharma Professional Research S.A. de C.V., Mexico City
  - Mexico Centre for Clinical Research S.A de C.V, Mexico City
  - Centro Estudios Clínicos y Esp. Médicas SC CECEM, Nuevo León
  - BIND Investigaciones S.C., San Luis Potosí City
  - Neurociencias Estudios Clinicos, Sinaloa
  - Centro para el Des de la Med y de Asist Med Esp SC, Sinaloa
- Serbia (13):
  - Clinical Hosp Center Dr Dragisa Misovic Dedinje, Belgrade
  - Clinical. Hospital Center Zvezdara, Belgrade
  - Institute of Mental Health, Belgrade
  - Special Hospital for Cerebrovascular Disease Sveti Sava, Belgrade
  - Special Hospital for Psychiatric Diseases, Gornja Toponica
  - Spl. Hosp. for Psychiatric Diseases Kovin, Kovin
  - Janjic University Clinical Center Kragujevac, Kragujevac
  - Jovanovic University Clinical Centre of Kragujevac, Kragujevac
  - University Clinical Center Kragujevac, Kragujevac
  - University Clinical Center Nis, Niš
  - Spl. Hosp. for Psychiatric Diseases Sveti Vracevi, Novi Kneževac
  - Gen. Hosp. Dr Radivoj Simonovic, Sombor
  - General Hospital Valjevo, Valjevo
- South Korea (8):
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Eunpyeong St. Mary's Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
- Spain (2):
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Provincial de Zamora, Zamora
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No